CLINICAL TRIAL: NCT00537277
Title: A Titrate-To-Target Study of the Efficacy and Safety of Biphasic Insulin Aspart 30 in Subjects With Type 2 Diabetes Mellitus Not Achieving Glycaemic Targets on OADs With / Without Once Daily Basal Insulin Therapy
Brief Title: Efficacy and Safety of Biphasic Insulin Aspart 30 in Type 2 Diabetes Mellitus When Failing on OADs
Acronym: IMPROVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1849
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Results first posted 2010-08-17 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIAsp 30 (Experimental): Biphasic insulin aspart 30 administered once daily for 16 weeks. If HbA1c is higher than 7.0 % after 16 weeks of treatment, dose is increased to twice daily for another 16 weeks. If HbA1c is higher than 7.0 % after 32 weeks of treatment, dose is increased to three times daily until week 48 (end of trial).
  Interventions: Drug: biphasic insulin aspart

INTERVENTIONS:
Drug: biphasic insulin aspart — Treat-to-target dose titration scheme (dose individually adjusted), injected s.c. (under the skin)
  Other Names: BIasp; NovoLog Mix 70/30; NovoMix 30

SUMMARY:
This trial is conducted in Europe.

This is a clinical trial investigating the effectiveness and the safety of using biphasic insulin aspart 30 both for initiation and intensification of insulin treatment in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus for more than 12 months
* HbA1c: 7.5 - 11.0%
* An antidiabetic regimen that has been stable for at least 3 months prior to screening
* An antidiabetic regimen that includes a minimum of 2 oral anti-diabetic drugs (OADs) or 1 OAD plus evening or bedtime basal insulin
* OADs dosed at 50% or more of the maximum recommended dose

Exclusion Criteria:

* Use of any insulin preparations other than NPH or glargine within the past 6 months
* Use of more than 60 units of insulin per day
* Morning time insulin administration
* Use of more than one insulin dose daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2007-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One single site in Turkey
Pre-assignment Details: Eligible subjects were those with type 2 diabetes inadequately controlled with oral anti-diabetic drugs (OADs) with or without basal insulin therapy.
Groups:
- BIAsp 30: Subjects received individually adjusted dose of biphasic insulin aspart 30 (BIAsp 30) once daily for 16 weeks. If the treatment target of HbA1c below 7% was reached after 16 weeks of treatment, the subject continued the reached dose until week 48 (end of trial). If the treatment target of HbA1c below 7% was not achieved at week 16, then BIAsp 30 treatment was increased to twice daily for additional 16 weeks. If the treatment target of HbA1c below 7% was reached after 32 weeks of treatment, the subject continued the reached dose until week 48 (end of trial). If the treatment target of HbA1c below 7% was not achieved at week 32, then BIAsp 30 treatment was increased to three times daily for additional 16 weeks until week 48 (end of trial).
Period: Overall Study
Arm/Group | BIAsp 30
Started | 161
Exposed to Trial Drug | 160 (One subject not exposed to trial drug, and thus not included in full analysis set (FAS))
Completed | 112
Not Completed | 49
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 12
Not completed — Protocol Violation | 11
Not completed — Unclassified | 4
Not completed — Inability to tolerate trial medication | 4
Not completed — Non-compliance with trial procedures | 15

BASELINE CHARACTERISTICS:
Arm/Group | BIAsp 30
Number analyzed (Participants) | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 62
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index
  kg/m^2 | 31.1 (5.7)
Diabetes Duration [Mean (Standard Deviation); unit: years] — Number of years since diagnosis
  years | 9.5 (5.1)
Height [Mean (Standard Deviation); unit: cm] | 161 (9.00)
Weight [Mean (Standard Deviation); unit: kg] | 80.2 (15.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving the Treatment Target of Glycosylated Haemoglobin (HbA1c) Below 7.0%
Time Frame: week 48
Population: Full Analysis Set (FAS) was all subjects who have been exposed to at least one dose of trial drug.
Measure: Number; unit: percentage of subjects
Arm/Group | BIAsp 30
Number analyzed (Participants) | 160
percentage of subjects
  Achieving treatment target HbA1c < 7.0% | 34.4
  Not achieving treatment target HbA1c < 7.0% | 46.9

2. Secondary Outcome: Percentage of Trial Completers Achieving the Treatment Target of Glycosylated Haemoglobin (HbA1c) Below 7.0%
Time Frame: week 48
Population: Full Analysis Set (FAS) was all subjects who have been exposed to at least one dose of trial drug.
Measure: Number; unit: percentage of trial completers
Arm/Group | BIAsp 30
Number analyzed (Participants) | 112
percentage of trial completers
  Achieving treatment target HbA1c < 7.0% | 48.2
  Not achieving treatment target HbA1c < 7.0% | 51.8

3. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: Total number of hypoglycaemic episodes experienced from baseline (week 0) to end of trial (week 48). Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose (PG) below 3.1 mmol/L or 56 mg/dL. Symptoms only if subject was able to treat her/himself and with either no PG or blood glucose measurement or PG higher than or equal to 3.1 mmol/L or 56 mg/dL.
Time Frame: weeks 0-48
Population: Safety analysis set was all subjects who have been exposed to at least one dose of trial drug.
Measure: Number; unit: episodes
Arm/Group | BIAsp 30
Number analyzed (Participants) | 160
episodes
  Major | 4
  Minor | 43
  Symptom only | 15

4. Secondary Outcome: Number of Diurnal Hypoglycaemic Episodes
Description: Total number of hypoglycaemic episodes during the day (diurnal) experienced in the trial from baseline (week 0) to end of trial (week 48). Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose (PG) below 3.1 mmol/L or 56 mg/dL. Symptoms only if subject was able to treat her/himself and with either no PG or blood glucose measurement or PG higher than or equal to 3.1 mmol/L or 56 mg/dL.
Time Frame: weeks 0-48
Population: Safety analysis set was all subjects who have been exposed to at least one dose of trial drug.
Measure: Number; unit: episodes
Arm/Group | BIAsp 30
Number analyzed (Participants) | 160
episodes
  Major | 2
  Minor | 33
  Symptom only | 13

5. Secondary Outcome: Number of Nocturnal Hypoglycaemic Episodes
Description: Total number of hypoglycaemic episodes during the night (nocturnal) experienced in the trial from baseline (week 0) to end of trial (week 48). Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose (PG) below 3.1 mmol/L or 56 mg/dL. Symptoms only if subject was able to treat her/himself and with either no PG or blood glucose measurement or PG higher than or equal to 3.1 mmol/L or 56 mg/dL.
Time Frame: weeks 0-48
Population: Safety analysis set was all subjects who have been exposed to at least one dose of trial drug.
Measure: Number; unit: episodes
Arm/Group | BIAsp 30
Number analyzed (Participants) | 160
episodes
  Major | 2
  Minor | 10
  Symptom only | 2

6. Secondary Outcome: Number of Treatment Emergent Serious Adverse Events (SAEs)
Description: Total number of treatment emergent SAEs experienced from baseline (week 0) to end of trial (week 48). A treatment emergent SAE were defined as an adverse event which occurred in the trial treatment period.
Time Frame: weeks 0-48
Population: Safety analysis set was all subjects who have been exposed to at least one dose of trial drug.
Measure: Number; unit: events
Arm/Group | BIAsp 30
Number analyzed (Participants) | 160
events | 7

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a time span of 48 weeks.
Description: Safety analysis set were all subjects who have been exposed to at least one dose of trial drug.
Arm/Group | BIAsp 30
Serious Adverse Events (participants affected / at risk) | 5/160
Other Adverse Events (participants affected / at risk) | 44/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 30 (N=160)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 30 (N=160)
Blood cholesterol increased (Investigations) | 11 (16)
Blood potassium increased (Investigations) | 8 (12)
Blood triglycerides increased (Investigations) | 13 (18)
Low density lipoprotein increased (Investigations) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk acknowledges the Investigator's right to publish the entire results of the trial. Any such scientific paper, presentation, communication or other information concerning the investigation described in this protocol, must be submitted in writing to Novo Nordisk Trial Manager prior to submission for publication/presentation for comments. Comments will be given within four weeks from receipt of the manuscript.